CLINICAL TRIAL: NCT02113774
Title: The Impact of Antimicrobial Treatment for Asymptomatic Bacteriuria in Renal Transplant Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Ruth Rahamimov, head of transplant investigator service, Rabin Medical Center
Purpose: Treatment
Other Study IDs: 7687
Record Dates: First submitted 2014-03-23; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Urinary Tract Infection; Bacteriuria; Renal Transplantation
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria

ARMS (2):
- no therapy (No Intervention)
- antimicrobial treatment according to in-vitro susceptibility (Active Comparator)
  Interventions: Other: antimicrobial treatment according to in-vitro susceptibility

INTERVENTIONS:
Other: antimicrobial treatment according to in-vitro susceptibility
  Arms: antimicrobial treatment according to in-vitro susceptibility

SUMMARY:
The investigators hypothesize that antibiotic therapy for asymptomatic bacteriuria in renal transplant patients does not have impact on the development of symptomatic urinary tract infection (UTI) or progression of renal impairment in patients during the first year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥1 month and ≤ 12 months after renal transplantation.
* Positive urine culture defined as ≥ 105 colony forming units (CFU) per milliliter of a known single pathogen.

Exclusion Criteria:

* Any one of the following signs and symptoms: fever, abdominal pain, dysuria, frequency, urgency, flank pain, costovertebral-angel tenderness or tenderness over the transplanted kidney
* Active infections in another site
* Leucocytosis (WBC >18.000K/micl) or leucopenia (WBC < 3.000 K/micl)
* Elevation of serum creatinine of more than 15% of its baseline level
* Obstructive or other urological complications following transplantation as known foreign device (stent/double-J-Cath, any catheter) in the urinary tract system, known obstruction of the transplanted kidney, indwelling or intermittent catheterization
* Pregnant or lactating women.
* Candidates to invasive urologic procedures.
* Inability to return for regular follow up.
* Previous enrollment in this study.
* Patients who incapable of giving informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2014-04; Primary Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
development of symptomatic urinary tract infection | 30 days

SECONDARY OUTCOMES:
25% reduction in estimated glomerular filtration rate (eGFR) | 1 year

OTHER OUTCOMES:
graft loss | 1 year